CLINICAL TRIAL: NCT05960019
Title: A Study of the Hypoglycemic Effect of African Traditional Fermented Foods Amongst Pre-diabetic Adults.
Brief Title: Blood Glucose Control Using African Traditional Fermented Foods
Acronym: ATFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Linnaeus University (Other); Kenyatta University (Other)
Responsible Party: Principal Investigator, Rosebella Iseme-Ondiek, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-104
Record Dates: First submitted 2023-04-19; First posted 2023-07-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fermented milk product (Experimental): Dietary supplement (Maziwa Mala) This is a type of cultured dairy milk, that is prepared through mesophilic fermentation of milk that is widely available in Kenya. Participants will be expected to consume 250ml of the mala each day for breakfast.
  Interventions: Dietary Supplement: Fermented milk product
- Fermented cereal based porridge (Experimental): Dietary supplement (Uji) This is a fermented cereal-based porridge prepared from a mix of ground millet and sorghum that is mixed with water into a gruel which is fermented into a non-alcoholic beverage or meal depending on desired thickness. Participants will be expected to consume 250ml of the porridge each day for breakfast.
  Interventions: Dietary Supplement: Fermented cereal based product
- Standard of Care (Active Comparator): Standard of care shall comprise behavioural (lifestyle) modification counselling delivered monthly. This shall consist of provision of counselling on lifestyle modification in an effort to help the participants prevent progression of the pre-diabetes and provide help with any emerging complications of the disease. Counselling on lifestyle modification shall comprise provision of standard dietary and exercise advice for pre-diabetics by a study doctor.
  Interventions: Behavioral: Behavioural modification counselling

INTERVENTIONS:
Dietary Supplement: Fermented milk product — This is a type of cultured bovine milk, that is prepared through mesophilic fermentation of milk, that is widely available in Kenya. Participants will be expected to consume 250ml of the mala each day for breakfast.
  Other Names: Maziwa mala
  Arms: Fermented milk product
Dietary Supplement: Fermented cereal based product — This is a fermented cereal-based porridge prepared from a mix of ground millet and sorghum that is mixed with water into a gruel which is fermented into a non-alcoholic beverage or meal depending on desired thickness. Participants will be expected to consume 250ml of the porridge each day for breakfast.
  Other Names: Uji
  Arms: Fermented cereal based porridge
Behavioral: Behavioural modification counselling — Standard of care shall comprise behavioural (lifestyle) modification counselling delivered monthly. This shall consist of provision of counselling on lifestyle modification in an effort to help the patients prevent progression of the pre-diabetes and provide help with any emerging complications of the disease. Counselling on lifestyle modification shall comprise provision of standard dietary and exercise advice for pre-diabetics by a study doctor.
  Other Names: Lifestyle modification counselling
  Arms: Standard of Care

SUMMARY:
Although African traditional fermented foods have been linked to health benefits, research pertaining to the use of uniform products in the control of blood glucose is lacking. This study is aimed at assessing the effectiveness of African traditional fermented foods at reducing blood sugar amongst adult pre-diabetic patients. This study shall comprise a multi-centre parallel (3-arm) randomized controlled trial of a fermented milk product, a fermented cereal-based product, and standard medical care. 252 pre-diabetic adults shall be recruited from 12 treatment facilities located at 4 Counties (3 clinics from each County) across Kenya. The primary outcome is change in glycated haemoglobin. Secondary outcomes shall include, change in weight (BMI), waist circumference, levels of fasting plasma glucose, C reactive protein and lipid profile. Safety as well as the acceptability and experience of fermented foods as a treatment modality for pre-diabetes will additionally be assessed amongst study participants. At each study site, data comprising clinical measurements and responses from self-report questionnaires shall be collected over a follow-up period of 12 weeks. Two focus group discussions shall additionally be held in week 13. Comparison of the mean changes between the three groups shall be carried out using Analysis of Variance (ANOVA). Pairwise comparisons shall additionally be undertaken using linear mixed regression models.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed pre-diabetes (diagnosed less than 6 months ago), defined as HbA1c between 5.7% and 6.4%,
* Both male and female prediabetic individuals
* Aged between 18 and 65 years
* Seeking clinic services at the selected AKU-outreach facilities for at least 3 visits (including seeking services for separate reasons other than pre-diabetes for the purpose of determining affiliation)

Exclusion Criteria:

* Currently on any of the following:

  * glucose lowering medication (including insulin therapy)
  * steroid therapy,
  * immunosuppressive therapy,
  * medication for gastric disease,
  * warfarin or other coumarin derivates,
  * Vitamin C or E, Iron or B12
  * erythropoietin
  * antiretrovirals
  * ribavirin
  * dapsone
* Chronic use (defined as consumption of more than 3 months) of non-steroidal anti-inflammatory drugs or aspirin
* Individuals that have consumed antibiotics in the last month.
* Individuals that regularly consume fermented foods or took nutritional supplements including probiotics during the 3 months prior to screening. Regular consumption shall be defined as consuming at least 250ml of fermented foods on six days in a week.
* Individuals who at the time of enrolment are smokers, regularly consume alcohol (defined as having had at least 12 drinks in the past year but 3 drinks or fewer per week, on average over the past year) or are suffering from drug addiction including chronic opiate use.
* Individuals with a history of gastrointestinal surgery (gastrectomy, bariatric surgery, or colostomy), splenectomy or gastrointestinal malignancy.
* Individuals known to be:

  * HIV+ve,
  * suffering from blood disorders such as Reticulocytosis or any form of Anaemia (including Iron deficiency, B12 Deficiency) or Haemoglobinopathies.
  * Pregnant or lactating,
  * with serious organic or metabolic conditions [such as malignant disease, pancreatitis, endocarditis, liver, or severe kidney disease (serum creatinine level above the normal range or macroalbuminuria including chronic renal failure), severe pulmonary or heart disease], splenomegaly, rheumatoid arthritis, hypertriglyceridemia, in a terminal stage of illness, or experiencing acute or severe episodes of mental illness at the time of enrolment.
* Individuals with allergies to dairy or cereal products such as millet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | "12 weeks"
  Change in levels of glycated haemoglobin

SECONDARY OUTCOMES:
Change in lipid profile | "4 weeks" and "12 weeks"
  Change in levels of total cholesterol, triglycerides, HDL, LDL
Change in weight | "4 weeks" and "12 weeks"
  Change in weight
Change in CRP levels | "4 weeks" and "12 weeks"
  Change in levels of inflammatory marker C reactive protein
Change in waist circumference | "4 weeks" and "12 weeks"
  Change in waist circumference
Change in FBG | "4 weeks" and "12 weeks"
  Change in levels of fasting blood glucose

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | "from date of randomization through to study completion, an average of 12 weeks"
  Adverse events occurring due to consumption of allocated fermented food

CONTACTS AND LOCATIONS:
Overall Officials: Rosebella A Iseme-Ondiek, PhD, Principal Investigator — Aga Khan University
Locations (2):
- Kenya (2):
  - Aga Khan Outreach Facilities, Kiambu
  - Aga Khan Outreach Facilities, Nairobi